CLINICAL TRIAL: NCT01944384
Title: Impacts of Aldosterone Blockade on Myocardial Remodeling in Hypertensive Patients With Diastolic Failing Heart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200912097M
Record Dates: First submitted 2013-09-04; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- aldactone (Experimental): aldactone 25 mg for 6 months
  Interventions: Drug: aldactone
- without aldactone (No Intervention)

INTERVENTIONS:
Drug: aldactone — aldactone 25 mg for 6 months
  Arms: aldactone

SUMMARY:
Aim of study: The effects of aldosterone blockade on myocardial remodeling in hypertensive patients with diastolic failing heart remains unclarified.

Background: Nearly half of patients with clinical heart failure (HF) have normal left ventricular ejection fraction (LVEF) who usually present with apparent diastolic dysfunction (DD) and are referred as diastolic HF (DHF). The renin-angiotensin-aldosterone system is an established major pathway that is operative in the pathogenesis of HF. The effects of aldosterone on myocardial hypertrophy, fibrosis and endothelial dysfunction have clearly been established in human and animal models. Furthermore, in these models, aldosterone antagonism prevented the development of myocardial fibrosis independent of its effect on blood pressure or myocardial hypertrophy. However, its application to patients with DHF is unspecified. In the study, we hypothesize that aldosterone blockade could reverse LV remodeling process in hypertensive patients with DHF.

Study protocol: We will enroll medically well-controlled hypertensive patients who have DHF defined as the presence of exertional dyspnea or HF signs/symptoms, diastolic dysfunction as impaired tissue-Doppler (TDI) derived mitral early annular diastolic velocity (< 8 cm/s), and LVEF > 50 % in echocardiography. All patients will be randomized to receive spironolactone 25 mg per day or not for at least 6 months. At baseline before randomization and 6 months after randomization, we will investigate the Quality-of-life (QOL) score by Minnesota Living with Heart Failure questionnaire (Chinese version), echocardiography coupled with TDI to assess the degree of LV hypertrophy, myocardial systolic and diastolic characteristics. Otherwise, we draw blood sampling at baseline and after randomization for quantifying and comparing several biomarkers which are currently proved to be correlated with LV hypertrophy, myocardial fibrosis, and biomechanical stretch in DHF patients, such as N-terminal pro-brain-type natriuretic peptide, matrix metalloproteinase-2, carboxy-terminal telopeptide, procollagen type III amino-terminal propeptide, soluble ST2, and galectin-3. Expected results: Aldosterone antagonism is effective for hypertensive patients with DHF by improving the quality of life, echo-derived myocardial function, and reducing ventricular mechanical stretch through lessening the degree of LV hypertrophy and myocardial fibrosis.

DETAILED DESCRIPTION:
Aim of study: The effects of aldosterone blockade on myocardial remodeling in hypertensive patients with diastolic failing heart remains unclarified. Background: Nearly half of patients with clinical heart failure (HF) have normal left ventricular ejection fraction (LVEF) who usually present with apparent diastolic dysfunction (DD) and are referred as diastolic HF (DHF). Hypertensive heart disease occurs in the majority of patients with DHF, and several key aspects of heart failure secondary to hypertensive heart disease are the relatively highly prevalent LV hypertrophy, cardiac fibrosis, and endothelial dysfunction-mediated myocardial injury caused by changes in the local and systemic neurohormonal environment, and all of which are associated with LV diastolic dysfunction and tissue-Doppler derived systolic myocardial function. The renin-angiotensin-aldosterone system is an established major pathway that is operative in the pathogenesis of HF. The effects of aldosterone on myocardial hypertrophy, fibrosis and endothelial dysfunction have clearly been established in human and animal models. Furthermore, in these models, aldosterone antagonism prevented the development of myocardial fibrosis independent of its effect on blood pressure or myocardial hypertrophy. However, its application to patients with DHF is unspecified. In the study, we hypothesize that aldosterone blockade could reverse LV remodeling process in hypertensive patients with DHF.

Study protocol: We will enroll medically well-controlled hypertensive patients who have DHF defined as the presence of exertional dyspnea or HF signs/symptoms, diastolic dysfunction as impaired tissue-Doppler (TDI) derived mitral early annular diastolic velocity (< 8 cm/s), and LVEF > 50 % in echocardiography. All patients will be randomized to receive spironolactone 25 mg per day or not for at least 6 months. At baseline before randomization and 6 months after randomization, we will investigate the Quality-of-life (QOL) score by Minnesota Living with Heart Failure questionnaire (Chinese version), echocardiography coupled with TDI to assess the degree of LV hypertrophy, myocardial systolic and diastolic characteristics. Otherwise, we draw blood sampling at baseline and after randomization for quantifying and comparing several biomarkers which are currently proved to be correlated with LV hypertrophy, myocardial fibrosis, and biomechanical stretch in DHF patients, such as N-terminal pro-brain-type natriuretic peptide, matrix metalloproteinase-2, carboxy-terminal telopeptide, procollagen type III amino-terminal propeptide, soluble ST2, and galectin-3. Expected results: Aldosterone antagonism is effective for hypertensive patients with DHF by improving the quality of life, echo-derived myocardial function, and reducing ventricular mechanical stretch through lessening the degree of LV hypertrophy and myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* well-controlled hypertensive patients with diastolic HF defined as the presence of diastolic dysfunction, normal LVEF (> 50 %), and exertional dyspnea (≧ New York Heart Association functional class II) or other HF signs/symptoms fulfilled with the Framingham criteria despite optimal pharmacological therapy

Exclusion Criteria:

* secondary hypertension
* restrictive, constrictive or hypertrophic cardiomyopathy
* more than moderate (mitral or tricuspid regurgitant jet area/atrial area more than 20%; aortic regurgitant jet to the tip of the mitral valve leaflets) valvular heart diseases
* chronic atrial fibrillation
* usage of aldosterone antagonist within 3 months
* chronic pulmonary disease
* myocardial infarction within 3 months or active ischemia needing revascularization
* LVEF less than 50% by echocardiography
* renal failure (serum creatinine concentration more than 2.0 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
peak myocardial velocity (Sm) during the ejection phase over the 6-basal segments | 6 months

SECONDARY OUTCOMES:
pro-brain natriuretic peptide (proBNP) | 6 months
matrix metalloproteinase-2 (MMP-2) | 6 months
matrix metalloproteinase-9 (MMP-9), etc. | 6 months
carboxy-terminal telopeptide of collagen I(ICTP) | 6 months
procollagen type III amino-terminal propeptide (PIIINP) | 6 months
soluble ST2 receptor (sST2) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yi Chih, MD, PhD, Principal Investigator — NTUH